CLINICAL TRIAL: NCT00201162
Title: Soy and Lipoproteins in Postmenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 280; R01HL070553 (NIH); NCT00181103 (obsolete NCT alias)
Record Dates: First submitted 2005-09-16; First posted 2005-09-20 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Atherosclerosis; Cardiovascular Diseases; Heart Diseases; Menopause
MeSH Terms: conditions — Atherosclerosis; Cardiovascular Diseases; Heart Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): dietary supplement soy protein containing isoflavones
  Interventions: Dietary Supplement: Soy
- Placebo (Placebo Comparator): dietary supplement casein placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Soy — Dietary supplement of isolated soy protein containing isoflavones
  Arms: Intervention
Dietary Supplement: Placebo — dietary supplement casein placebo
  Arms: Placebo

SUMMARY:
To determine the effects of soy on lipids, lipoproteins and lipoprotein subclass in a sample of African-American and white postmenopausal women with low-density lipoprotein (LDL) cholesterol elevations that may increase their lifetime risk for cardiovascular disease but would not qualify for definite pharmacotherapy under current guidelines.

DETAILED DESCRIPTION:
BACKGROUND:

Cardiovascular disease (CVD) remains the leading cause of mortality and disability in postmenopausal women. Menopause alters serum lipids and lipoproteins to produce a more atherogenic lipid profile that may contribute significantly to the increased risk for the development of CVD over the lifetime of women. Clinical trials have demonstrated a beneficial effect of soy protein containing isoflavones (soy) on plasma lipids and lipoproteins; however, these studies included small numbers of postmenopausal women and virtually none included sufficient African-American women. In addition, no published data existed in 2001 on the impact of soy on atherogenic lipoprotein subclasses in postmenopausal women.

DESIGN NARRATIVE:

The study was a double blind, parallel group, randomized clinical trial. A total of 216 healthy postmenopausal women (50 percent African-American) with LDL cholesterol between 130 mg/dL and 190 mg/dL were enrolled. Following a pre-randomization run-in period on a NCEP Step I diet, women were randomized to receive soy containing isoflavones or casein dietary supplements for 3 months. Major outcome variables were assessed in both groups at baseline and again at 3 months. It was hypothesized that soy supplementation would result in significantly greater reduction in LDL cholesterol, LDL particle concentration, and prevalence of dense LDL particles and improvement in menopausal quality of life compared with placebo and that these effects would be comparable in African-Americans and whites. This was the first study to determine whether a natural plant product could ameliorate the unfavorable changes in known and novel lipid risk factors that are a consequence of menopause in both African-American and white women. The unique transitional outcomes explored in this study added substantially to the limited body of knowledge of the effects of soy. Evaluation of this nutritional alternative to hormone replacement therapy (HRT) that may provide a beneficial effect on lipid risk factors and menopausal symptoms but would be free of the adverse effects on triglycerides, the breast and uterus, and thrombotic events associated with HRT could have significant public health implications for postmenopausal women.

ELIGIBILITY:
Inclusion criteria

* postmenopausal women
* elevated cholesterol

Ages: 50 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2001-09; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
LDL cholesterol level | 3 months
  LDL cholesterol will be measured in blood in mg/dl

CONTACTS AND LOCATIONS:
Overall Officials: Jerilyn Allen, Principal Investigator — Johns Hopkins University